CLINICAL TRIAL: NCT01931540
Title: Developmental ORIgins of Healthy and Unhealthy AgeiNg: the Role of Maternal Obesity
Acronym: DORIAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other); University of Helsinki (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); Istituto Superiore di Sanità (Other)
Responsible Party: Principal Investigator, Pirjo Nuutila, MD PhD, Turku University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T55/2012b; EC-FP7-278603 (Other Grant/Funding Number: EC within the FP7 under the project DORIAN, GA n° 278603)
Record Dates: First submitted 2013-04-22; First posted 2013-08-29 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Maternal-Fetal Relations; Muscle Weakness; Insulin Resistance
Keywords: Obesity; Epigenesis, Genetic; Exercise Therapy
MeSH Terms: conditions — Muscle Weakness; Insulin Resistance; Obesity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise Training - 17 offspring of OM (Experimental): 4 months exercise training, OM: Obese mothers
  Interventions: Behavioral: Exercise Training
- 11 non-frail controls (9 LM) (No Intervention): Studied only at baseline
- Exercise Training - 20 offspring of LM (Experimental): 4 months exercise training, LM:Lean/Normal Mothers
  Interventions: Behavioral: Exercise Training

INTERVENTIONS:
Behavioral: Exercise Training — Three times a week, for four months.
  Arms: Exercise Training - 17 offspring of OM; Exercise Training - 20 offspring of LM

SUMMARY:
The prevalence of obesity in the developed world has increased markedly over the last 20 years. Considering the prevalence of obese and overweight adult subjects, and the fact that pregnancy itself induces a state of insulin resistance and inflammation, maternal obesity may be the most common health risk for the developing fetus. It is well established that what we eat has a major impact on our health. However, there is growing evidence to suggest that diet during pregnancy and lactation may be particularly important as not only does it influence the health of the mother, it may have a permanent effect on the health of her children and even her grandchildren. The concept that environmental factors, such as nutrition during early development, influence both our health span and lifespan has been termed the developmental origins of health and disease hypothesis.

The objective of the study are:

* to compare subjects with frailty (condition developed with ageing) with controls and characterize the unhealthy aged condition with the measurements described below
* to examine if signs of frailty can be reversed by lifestyle induced modifications (exercise training programme) of its primary components (IR, sarcopenia, psychological profile) in offspring of overweight/obese (OOM) vs lean mothers (OLM).

The study consists of 37 frail old subjects, age ≥ 65 sub-grouped in 17 OOM, and 20 OLM and 11 non frail controls. These subjects will be studied with positron emission tomography (PET), computed tomography (CT), magnetic resonance imaging (MRI) and spectroscopy (MRS) and ultra sounds (US). In addition functional MRI (fMRI) will be performed. Adipose tissue biopsies will be taken.

Subjects will undergo characterization of biohumoral markers, a 75 g oral glucose tolerance test, imaging biomarkers (PET/CT, US, fMRI-MRS), genetic biomarkers (DNA and telomere damage) and inflammatory biomarkers (macrophage infiltration) before and after the 4-month lifestyle intervention period (physical exercise). By PET/CT it will be measured tissue-specific IR in skeletal muscle, adipose tissue, liver, myocardium and targeted brain regions. MRS will be used to measure organ steatosis in the skeletal muscle and liver, MRI will be used to measure fat masses in abdominal areas, and fMRI will be performed to assess activation in brain regions regulating cognition and appetite/energy control. US will be used to assess cardiovascular markers (IMT, strain and function).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be already participating the Helsinki Birth Cohort Study

Frailty Groups Inclusion Criteria:

* (Frailty) with lowest half of adult grip strength (measured 2001-2004)
* Group OM: (Offspring of Obese mothers) Highest quartile of maternal BMI
* Group LM: (Offspring of Normal weight/Lean mothers) Lowest two quartiles of maternal BMI

Control group Inclusion Criteria:

* (no Frailty) with highest half of adult grip strength (measured 2001-2004)
* Offspring of normal weight mothers

Exclusion Criteria:

* Subjects whose mothers were pre-eclamptic during pregnancy
* Oral corticosteroid or Warfarin therapy
* Recent myocardial infarction
* Severe chronic disorder that can prevent to participate the intervention
* Chronic atrial fibrillation and pacemaker
* Cancer less than 5 years ago
* Current smoking
* Diabetes requiring insulin treatment or fasting glucose more than 7 mmol/l
* Weight more than 170 kg and Waist circumference > 150 cm
* Inner ear implants
* Metal objects in body including metallic prostheses, artificial valve prostheses, surgical clips, braces, foreign fragments or tattoo

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Baseline group comparison and Change from Baseline in Insulin-stimulated whole body and organ-specific glucose uptake at 4 months | At day 1 and after 4 months of intervention (for the 15 controls only at baseline)
  Assessed via 18F-Fluorodeoxyglucose (FDG)-PET/CT+Clamp technique
Baseline group comparison and Change from Baseline in Epigenetic characterization of DNA samples (Telomere length, H2A.X phosphorilation, mtDNA deletion, p66) at 4 months | At day 1 and after 4 months of intervention (for the 15 controls only at baseline)
  Telomere length, H2A.X phosphorilation, mtDNA deletion are measurements performed in Pisa, National Research Council p66 presence is measured in Rome, Istituto Superiore di Sanita'

SECONDARY OUTCOMES:
Baseline group comparison and Change from Baseline in Fat masses and content via MRI and MRS at 4 months | At day 1 and after 4 months of intervention (for the 15 controls only at baseline)
  Adipose tissue fat masses in different depots (subcutaneous, visceral, pericardial) Liver, skeletal muscle, vertebral fat content
Baseline group comparison and Change from Baseline in MRI brain anatomy and fMRI characterization of activation response to food stimuli of different brain regions at 4 months | At day 1 and after 4 months of intervention
  MRI anatomy: White matter volume, Cortex thickness, Nerve tracks found with Diffusor Tension Imaging fMRI will be used to identify different brain regions activated by food stimuli while subjects perform three different task: watch the food, think of eating the food, control the urge to eat the food.

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, MD PhD, Principal Investigator — Turku PET Centre (Turku University Hospital)
Locations (2):
- Finland (2):
  - University of Helsinki, Department of General Practice and Primary Health Care, Helsinki
  - Turku PET Centre (Turku University Hospital), Turku

REFERENCES:
- [Derived] Berry A, Bucci M, Raggi C, Eriksson JG, Guzzardi MA, Nuutila P, Huovinen V, Iozzo P, Cirulli F. Dynamic changes in p66Shc mRNA expression in peripheral blood mononuclear cells following resistance training intervention in old frail women born to obese mothers: a pilot study. Aging Clin Exp Res. 2018 Jul;30(7):871-876. doi: 10.1007/s40520-017-0834-4. Epub 2017 Sep 26. PMID 28952131
- [Derived] Huovinen V, Bucci M, Lipponen H, Kiviranta R, Sandboge S, Raiko J, Koskinen S, Koskensalo K, Eriksson JG, Parkkola R, Iozzo P, Nuutila P. Femoral Bone Marrow Insulin Sensitivity Is Increased by Resistance Training in Elderly Female Offspring of Overweight and Obese Mothers. PLoS One. 2016 Sep 26;11(9):e0163723. doi: 10.1371/journal.pone.0163723. eCollection 2016. PMID 27669153
- [Derived] Bucci M, Huovinen V, Guzzardi MA, Koskinen S, Raiko JR, Lipponen H, Ahsan S, Badeau RM, Honka MJ, Koffert J, Savisto N, Salonen MK, Andersson J, Kullberg J, Sandboge S, Iozzo P, Eriksson JG, Nuutila P. Resistance training improves skeletal muscle insulin sensitivity in elderly offspring of overweight and obese mothers. Diabetologia. 2016 Jan;59(1):77-86. doi: 10.1007/s00125-015-3780-8. PMID 26486356